CLINICAL TRIAL: NCT03786744
Title: Efficiency Evaluation of Allogenic Umbilical Cord Blood (UCB) Transfusion in Patients With Autism
Brief Title: Allogenic Cord Blood Transfusion in Patients With Autism
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: State-Financed Health Facility "Samara Regional Medical Center Dinasty" (Other)
Responsible Party: Principal Investigator, Volchkov Stanislav, Deputy director, Quality assurance director, State-Financed Health Facility "Samara Regional Medical Center Dinasty"
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12112018
Record Dates: First submitted 2018-12-21; First posted 2018-12-26 (Actual); Results first posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-10

CONDITIONS: Autism Spectrum Disorder; Autism
Keywords: Autism, ASD, Cord blood
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This is prospective, non-randomized (open label) with control group study. The total 20 patient will be enrolled in this study. In 10 patient with ASD will be infused with umbilical corb blood. Other 10 patient with ASD will be treated with standard therapy (control group).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASD CB-MNC injection. (Experimental): ASD CB-MNC injection from different donors and standard therapy.
  Interventions: Biological: ASD CB-MNC injection.; Other: Standard therapy.
- Standard therapy. (Other): Patients with standard therapy as control group.
  Interventions: Other: Standard therapy.

INTERVENTIONS:
Biological: ASD CB-MNC injection. — CB-MNC injection from different donors. One dose consist 20-50 mil MNC/kg.The protocol include 3 injection at monthly intervals.
  Arms: ASD CB-MNC injection.
Other: Standard therapy. — The standard therapy can include drugs, special psychology training etc.

SUMMARY:
Autism is one of those disorders in Autism spectrum disorders (ASD), which characterized by social interaction abnormalities, impaired verbal and non-verbal communication, and repetitive, obsessive behavior, while the therapeutic effect of current treatments remains limited progress.

The possible reason for ASD is neural hypoperfusion and immune deregulation. The Human Umbilical Cord Blood Mononuclear Cells (hUCB-MNCs) have been shown to have the ability to modulate the immune response and enhance angiogenesis, suggesting the novel and promising therapeutic strategy. In this study, the safety and efficacy of hUCB-MNCs infusion will be evaluated in patients with Autism.

DETAILED DESCRIPTION:
Autism Spectrum Disorders (ASD) are heterogeneous neuro-developed disorders. Autism is the most common disorder of the diseases characterized by dysfunctions in response social interaction and communication, as well as the presence of repetitive and stereotyped behaviors. Recent reports of a sharp increase in the number of children with autism. The exact etiology of autism remains unclear. Compliance, the definition of effective treatments for autism is particularly difficult.

Although it has been understood, it can be a question of immune dysregulation. Examination of the inflammatory cytokines, dysfunction of the immune system and the immune system. The Human Umbilical Cord Blood Mononuclear Cells (hUCB-MNCs) have been shown to have the ability to modulate the immune response and enhance angiogenesis, suggesting the novel and promising therapeutic strategy. The Our study suggest that infusion of cord blood mononuclear cells will affect Autism.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis: autistic type disorder (ASD).
* Systemic speech underdevelopment
* The presence of attention deficit hyperactivity disorder as a comorbid state
* Cognitive impairment

Exclusion Criteria:

* organic pathology of the brain according to CT, MRI
* the presence of the following diseases in history: heart failure in the stage of decompensation, stroke in history less than 1 year ago, blood diseases;
* decompensation of chronic and endocrinological diseases;
* acute respiratory viral and bacterial infections, period less than 1 month after the acute phase.
* HIV infection, hepatitis B and C.
* oncological diseases, chemotherapy in the anamnesis;
* tuberculosis.
* Severe form of intellectual disability.
* Cerebral palsy.
* epilepsy.

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2018-10-12 (Actual); Primary Completion 2019-10-12 (Actual); Study Completion 2019-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: STANISLAV VOLCHKOV, MD, PhD, Principal Investigator — Medical Centre Dinasty
Locations (1):
- Medical Centre Dinasty, Samara, Russia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ASD CB-MNC Injection. | Standard Therapy.
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ASD CB-MNC Injection. | Standard Therapy. | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 10 | 20
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 7.95 [4.5 to 14] | 7.80 [4.3 to 13] | 7.87 [4.3 to 14]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 9 | 8 | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Russia | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: A Number of Participants With Non-serious and Serious Adverse Events 24 Hrs Post-transfusion
Description: Safety assessment. The adverse events rate will be assessed in all patients.
Time Frame: 24hrs post transfusion
Measure: Number; unit: participants
Groups:
- Control Group: The standard therapy can include drugs, special psychology training etc.
Arm/Group | ASD CB-MNC Injection. | Control Group
Number analyzed (Participants) | 10 | 10
participants
  Increase in body temperature | 0 | 0
  Chill | 0 | 0
  Hypotension | 0 | 0
  Dyspnea | 0 | 0
  Skin itching | 0 | 0
  Hives | 0 | 0
  Post-transfusion purple | 0 | 0
  Oedema Quinque | 0 | 0
  Oliguria | 0 | 0
  Hematuria | 0 | 0
  Jaundice | 0 | 0
  Nausea | 0 | 0
  Vomiting | 0 | 0
  Dizziness | 0 | 0
  Pain at injection site | 1 | 0
  Anxiety | 2 | 0

2. Primary Outcome: Autism Treatment Evaluation Checklist (ATEC).
Description: The ATEC is designed to measure changes in the severity of ASD in response to treatment. A total score and 4 subscale scores are reported. Questions in the first 3 subscales are scored using a 0-3 scale (not true/partially true/absolutely true). The 4 subscale, Health/Physical/Behavior, is scored using a 0-4 point scale (Not a problem/Minor problem/Moderate problem/Serious problem). The first subscale, Speech/Language/Communication, contains 14 items where the score ranges from 0-28 points. The Sociability subscale contains 20 items and participants can score from 0-40. The third subscale, Sensory/Cognitive awareness, has 18 items and scores range from 0-36. Finally, the Health/Physical/Behavior subscale contains 25 items and scores range from 0-75. The scores from each subscale are combined in order to calculate a Total Score, which ranges from 0 to179 points. A lower score indicates less severe symptoms of ASD and a higher score correlates with more severe symptoms of ASD.
Time Frame: score at baseline, 1, 2, 6, 12 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | ASD CB-MNC Injection. | Standard Therapy.
Number analyzed (Participants) | 10 | 10
score on a scale
  Speech/Language/Communication at baseline | 14 [10 to 20] | 14 [13 to 21]
  Speech/Language/Communication at 1 months | 11 [5 to 18] | 14 [11 to 21]
  Speech/Language/Communication at 2 months | 7 [2 to 17] | 16 [14 to 22]
  Speech/Language/Communication at 6 months | 11 [5 to 22] | 14 [12 to 20]
  Speech/Language/Communication at 12 months | 12 [6 to 17] | 15 [13 to 20]
  Sociability at baseline | 11 [9 to 17] | 11 [9 to 15]
  Sociability at 1 months | 11 [9 to 13] | 12 [9 to 15]
  Sociability at 2 months | 9 [6 to 14] | 11 [10 to 14]
  Sociability at 6 months | 11 [8 to 14] | 13 [10 to 15]
  Sociability at 12 months | 12 [8 to 14] | 14 [11 to 14]
  Sensory/Cognitive Awareness at baseline | 13 [9 to 14] | 12 [10 to 15]
  Sensory/Cognitive Awareness at 1 months | 10 [6 to 15] | 11 [10 to 17]
  Sensory/Cognitive Awareness at 2 months | 10 [5 to 11] | 11 [11 to 16]
  Sensory/Cognitive Awareness at 6 months | 12 [8 to 14] | 14 [11 to 16]
  Sensory/Cognitive Awareness at 12 months | 12 [7 to 13] | 13 [11 to 17]
  Health/ Physical Development/Behaviour at baseline | 24 [19 to 30] | 24 [19 to 30]
  Health/ Physical Development/Behaviour at 1 months | 16 [13 to 21] | 24 [19 to 30]
  Health/ Physical Development/Behaviour at 2 months | 14 [7 to 18] | 23 [19 to 30]
  Health/ Physical Development/Behaviour at 6 months | 16 [13 to 25] | 24 [19 to 30]
  Health/ Physical Development/Behaviour at 12months | 13 [10 to 17] | 22 [19 to 30]
  Total score at baseline | 63 [56 to 66] | 62 [59 to 73]
  Total score at 1 months | 55 [43 to 60] | 65 [60 to 72]
  Total score at 2 months | 44 [31 to 57] | 68 [59 to 76]
  Total score at 6 months | 55 [49 to 65] | 70 [60 to 82]
  Total score at 12 months | 55 [38 to 61] | 71 [60 to 81]
Statistical Analysis 1: Comparison: ASD CB-MNC Injection. vs Standard Therapy; The study results were statistically processed using parametric and non-parametric methods using STATA version 9.0, Statistica for Windows version 6.0. Changes from the beginning of therapy and after 1, 2, 6, 12 months were compared using the Wilcoxon criterion, data between the main group and the control group were compared using non-parametric method, Mann-Whitney test was used (data are presented in Me - median format with an indication of 25% and 75% quartile; Test type: Superiority; p = 0.049367, Wilcoxon (Mann-Whitney) — Alternative hypothesis: can be changed of speech, language, communication skills for Cord Blood versus Placebo groups in 2-month Threshold <0.05; Mean Difference (Net) = 9
Statistical Analysis 2: Comparison: ASD CB-MNC Injection; The study results were statistically processed using parametric and non-parametric methods using STATA version 9.0, Statistica for Windows version 6.0 and MS Office Excel 2007. Changes from the beginning of therapy and after 1, 2, 6, 12 months were compared using the Wilcoxon criterion, data between the main group and the control group were compared using non-parametric method, Mann-Whitney test was used (data are presented in Me - median format with an indication of 25% and 75% quartile; Test type: Superiority; p = 0.004072, Wilcoxon (Mann-Whitney) — Alternative hypothesis: can be changed average of 2-month of Health/Physical Development/Behaviour for Cord Blood versus Control groups. Threshold <0.05; Median Difference (Net) = 9
Statistical Analysis 3: Comparison: ASD CB-MNC Injection; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.017258, Wilcoxon (Mann-Whitney) — Alternative hypothesis: can be changed average of 12-month of Health/Physical Development/Behaviour for Cord Blood versus Placebo groups. Threshold <0.05; Mean Difference (Net) = 9
Statistical Analysis 4: Comparison: ASD CB-MNC Injection; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.031210, Wilcoxon (Mann-Whitney) — Alternative hypothesis: can be changed average of 1-month of total score for Cord Blood versus Placebo groups. Threshold <0.05; Mean Difference (Net) = 10
Statistical Analysis 5: Comparison: ASD CB-MNC Injection; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.001940, Wilcoxon (Mann-Whitney) — Alternative hypothesis: can be changed average of 2-month of Total score for Cord Blood versus Placebo groups. Threshold <0.05; Mean Difference (Net) = 24
Statistical Analysis 6: Comparison: ASD CB-MNC Injection; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.031210, Wilcoxon (Mann-Whitney) — Alternative hypothesis: can be changed average of 6-month of Total score for Cord Blood versus Placebo groups. Threshold <0.05; Mean Difference (Net) = 15
Statistical Analysis 7: Comparison: ASD CB-MNC Injection; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.011330, Wilcoxon (Mann-Whitney) — Alternative hypothesis: can be changed average of 12-month of Total score for Cord Blood versus Placebo groups. Threshold <0.05; Mean Difference (Net) = 16

3. Secondary Outcome: Cytokine Analysis.
Description: IL1b, IL6, TNF-alpha, IL8, y-IFN measure in patient peripheral blood
Time Frame: score at baseline, 1, 2, 6 months
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | ASD CB-MNC Injection.
Number analyzed (Participants) | 10
pg/mL
  y-IFN pg/ml at baseline | 0 [0 to 0]
  y-IFN pg/ml at 1 months | 0 [0 to 0]
  y-IFN pg/ml at 2 months | 0 [0 to 0]
  y-IFN pg/ml at 6 months | 0 [0 to 0]
  IL1b pg/ml at baseline | 1.228 [0 to 2.62]
  IL1b pg/ml at 1 months | 1.279 [0 to 3.117]
  IL1b pg/ml at 2 months | 1.9675 [0.095 to 3.251]
  IL1b pg/ml at 6 months | 2.794 [0.396 to 3.103]
  IL6 pg/ml at baseline | 1.0225 [0.43 to 2.168]
  IL6 pg/ml at 1 months | 0.673 [0.392 to 2.076]
  IL6 pg/ml at 2 months | 0.5625 [0.195 to 0.753]
  IL6pg/ml at 6 months | 0.7455 [0.494 to 0.863]
  IL8 pg/ml at baseline | 3.9175 [1.913 to 9.822]
  IL8 pg/ml at 1 months | 2.7985 [2.157 to 5.341]
  IL8 pg/ml at 2 months | 2.7485 [1.197 to 3.348]
  IL8 pg/ml at 6 months | 4.7975 [3.507 to 38.388]
  TNF-alpha pg/ml at baseline | 0 [0 to 0]
  TNF-alpha pg/ml at 1 months | 0 [0 to 0]
  TNF-alpha pg/ml at 2 months | 0 [0 to 0]
  TNF-alpha pg/ml at 6 months | 0.0 [0 to 0]

4. Secondary Outcome: Immune Status as Determined by Percentage of Peripheral Blood Cells
Description: Peripheral blood flow cytometry cell count for CD3; CD4; CD8; CD19; CD16-56 (%)
Time Frame: score at baseline, 6 month
Measure: Median (Inter-Quartile Range); unit: percentage of cells
Arm/Group | ASD CB-MNC Injection.
Number analyzed (Participants) | 10
percentage of cells
  CD 3+(%) at baseline | 61.24 [58.55 to 66.59]
  CD 3+(%) at 6 months | 63.71 [58.56 to 67.83]
  СD3+СD8+ (%) at baseline | 24.33 [22.36 to 25.58]
  СD3+СD8+(%) at 6 months | 25.345 [20.19 to 26.15]
  СD3+СD4+ (%) at baseline | 32.835 [29.14 to 36.3]
  СD3+СD4+(%) at 6 months | 32.55 [30.26 to 35.46]
  СD3+СD4+СD8+ (%) at baseline | 0.215 [0.19 to 0.25]
  СD3+СD4+СD8+(%) at 6 months | 0.31 [0.25 to 0.42]
  СD16+СD56+(%) at baseline | 15.19 [7.29 to 21.08]
  СD16+СD56+(%) at 6 months | 16.05 [11.47 to 21]
  СD19+(%) at baseline | 19.29 [17.46 to 21.67]
  СD19+ (%) at 6 months | 17.255 [16.25 to 18.68]

5. Secondary Outcome: Immune Status as Determined by Absolute Cell Count of Peripheral Blood Cells
Description: Peripheral blood flow cytometry cell count for CD3; CD4; CD8; CD19; CD16-56 (absolute v.)
Time Frame: score at baseline, 6 month
Measure: Median (Inter-Quartile Range); unit: cells/µl
Arm/Group | ASD CB-MNC Injection.
Number analyzed (Participants) | 10
cells/µl
  CD 3+ at baseline | 1450.355 [1364.77 to 2163.81]
  CD 3+at 6 months | 1829.11 [1507.34 to 2312.87]
  CD 3+CD8+ at baseline | 598.48 [481.48 to 790.19]
  CD 3+CD8+ at 6 months | 654.385 [600.56 to 819.81]
  CD 3+CD4+ at baseline | 750.08 [649.35 to 1197.94]
  CD 3+CD4+ at 6 months | 877.095 [752.35 to 1197.99]
  CD 3+ CD4+CD8+ at baseline | 5.555 [3.59 to 7.09]
  CD 3+ CD4+CD8+ at 6 months | 8.656 [7.46 to 10.93]
  CD 16+CD56+ at baseline | 321.89 [188.46 to 550.36]
  CD 16+CD56+ at 6 months | 476.055 [306.37 to 607.71]
  СD19+ at baseline | 457.505 [431.81 to 839.35]
  СD19+ at 6 months | 506.365 [392.8 to 650.88]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | ASD CB-MNC Injection. | Standard Therapy.
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 6/10 | 8/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ASD CB-MNC Injection. (N=10) | Standard Therapy. (N=10)
Infectious nature (Cardiac disorders) | 0 (0) | 0 (0)
Non Infectious nature (Cardiac disorders) | 0 (0) | 0 (0)
Infectious nature (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 4 (7) — 3 cases of influenza 1. case laryngitis 2. case tracheobronchitis
NON Infectious nature (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Infectious nature (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0)
NON Infectious nature (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Infectious nature (Renal and urinary disorders) | 0 (0) | 0 (0)
NON Infectious nature (Renal and urinary disorders) | 1 (1) | 0 (0)
Infectious nature (Gastrointestinal disorders) | 2 (2) | 1 (1) — food toxicology
NON Infectious nature (Gastrointestinal disorders) | 1 (1) | 2 (2) — Gastritis
Infectious nature (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0)
NON Infectious nature (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0)
Infectious nature (Nervous system disorders) | 0 (0) | 0 (0)
NON Infectious nature (Nervous system disorders) | 2 (3) | 1 (1) — head pain, dizziness
Psychiatric symptoms (Psychiatric disorders) | 1 (1) | 1 (1) — aggression irritability anxiety
Hypersensitivity (Immune system disorders) | 1 (1) | 2 (3) — seasonal allergy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-12): https://cdn.clinicaltrials.gov/large-docs/44/NCT03786744/Prot_SAP_000.pdf